CLINICAL TRIAL: NCT06598930
Title: Evaluation of the Efficacy of Intensive Medical Follow-up with an Advanced Practice Nurse Compared with Medical Follow-up Alone, in Non-severe Pulmonary Embolism - Randomised Open Study At Dijon University Hospital and Langres University Hospital.
Brief Title: Evaluation of the Effectiveness of Intensive Medical Follow-up with an Advanced Practice Nurse Compared with Medical Follow-up Alone in Non-severe Pulmonary Embolism.
Acronym: InCaPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANTEMI-RIBREUX AOIparaM 2023
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Non-severe Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive follow-up (Experimental)
  Interventions: Other: Intensive follow-up
- Routine follow-up (Active Comparator)
  Interventions: Other: Routine follow-up

INTERVENTIONS:
Other: Routine follow-up — As recommended: a vascular doctor exclusively, face-to-face consultations.
  Arms: Routine follow-up
Other: Intensive follow-up — a vascular physician and an IPA, with alternating face-to-face and remote consultations.
  Arms: Intensive follow-up

SUMMARY:
In France, venous thromboembolism (VTE), which includes pulmonary embolism (PE) and deep-vein thrombosis (DVT), is the 3rd leading cause of cardiovascular disease, leading to major public health problems. Despite current monitoring and treatment, the recurrence rate and the rate of haemorrhagic complications remain high, at 18.5% and 12% respectively in the year following the thrombotic event.

Patients with PE diagnosed in the emergency department are very often admitted to hospital.

However, according to international recommendations on the treatment of PE, outpatient management with early discharge could be envisaged but is rarely carried out in practice, particularly for non-severe PE (spESI = 0).

Current post-pulmonary embolism follow-up involves an early medical consultation with a specialist after discharge from hospital, with follow-up at 1, 3 and 6 months. The aim is to evaluate anticoagulant treatment (high-risk medication), investigate the causes of PE, monitor the patient and decide whether or not to continue anticoagulant treatment 6 months after diagnosis.

Patients diagnosed with non-severe PE can only be monitored as soon as they are discharged from hospital, thanks to an organised and specific care pathway involving healthcare professionals working in towns and cities as well as in hospitals.

In 2018, the French authorities created a new healthcare profession, the advanced practice nurse (APN). They are said to be one of the 'answers' to making care pathways, including PE, even more relevant by improving the quality of patient care and strengthening the town-hospital link.

Thanks to their training and expertise, IPAs can carry out the following activities:

* Observation, collection and interpretation of data in the context of patient monitoring in his/her area of expertise;
* Prescribing, renewing prescriptions and carrying out technical procedures as part of patient follow-up in their area of expertise;
* Designing, implementing and evaluating preventive and therapeutic education measures.

Thus, by intervening at specific times throughout the course of a patient's diagnosis of a non-severe PE, the involvement of the IPA in the patient's follow-up, in addition to current recommendations, would make it possible to reduce the risk of haemorrhagic complications associated with the use of anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given oral consent
* Person affiliated to the social security system
* Over 18 years of age
* Resident in the 21-52 region
* Emergency care at Dijon University Hospital or Langres University Hospital less than 24 hours after diagnosis of non-severe pulmonary embolism (spESI = 0)

Symptomatic PE is confirmed if there is :

* a high pre-test clinical probability and a high probability ventilation-perfusion (V/Q) lung scan according to the Prospective Investigation of Pulmonary Embolism Diagnosis (PIOPED) criteria
* a proximal DVT diagnosed by ultrasound in a patient with symptoms of PE;
* a positive CT pulmonary angiogram (PA) showing a central filling defect highlighted by contrast material or a complete occlusion in a segmental or more proximal pulmonary artery.
* No contraindication to anticoagulant treatment

Exclusion Criteria:

* Person not affiliated to or not benefiting from a social security scheme
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant women, women in labour or breastfeeding mothers
* An adult who is incapable or unable to give consent
* Minors
* Contraindication to anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of minor and major bleeds | Through study completion, on average of 7 months
  ISTH definition of haemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France